CLINICAL TRIAL: NCT03178968
Title: Can Surface Roughness Predict Progression of Tooth Wear in Participants With Dietary Origins of Acid?
Brief Title: Can Surface Roughness Predict Progression of Tooth Wear?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15/LO/0417
Record Dates: First submitted 2017-05-30; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Tooth Wear
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single-blind, randomised intervention study (blinded for the surface roughness measurements, step height measurements and microhardness testing)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 15 minutes' erosion (Experimental): Orange juice is administered ex vivo and in vivo for 5 minutes and repeated a total of 3 times
  Interventions: Other: Orange juice
- 30 minutes' erosion (Experimental): Orange juice is administered ex vivo and in vivo for 10 minutes and repeated a total of 3 times
  Interventions: Other: Orange juice
- 45 minutes' erosion (Experimental): Orange juice is administered ex vivo and in vivo for 15 minutes and repeated a total of 3 times
  Interventions: Other: Orange juice

INTERVENTIONS:
Other: Orange juice — 3 immersion times in orange juice were investigated

SUMMARY:
The clinical study was a single-blind, randomised intervention study to measure surface changes of polished and unpolished enamel in situ following an orange juice acid challenge. Ethical approval for the study was granted by the Stanmore Health Research Authority REC ref 15/LO/0417, and the study was conducted per the guidelines for Good Clinical Practice. The study investigated a total 6 erosion regimes divided in 3 different erosion times plus ex vivo immersion in orange juice drink versus in vivo rinsing of the same orange juice drink.

DETAILED DESCRIPTION:
60 unpolished and 60 polished enamel samples were prepared from extracted human molars collected under ethical approval.

30 healthy volunteers were recruited and lower dental impressions were recorded using standard stock trays. Custom made lower orthoodontic type appliances were made by the laboratory to accommodate a total of four enamel (2 left and right hand side) samples positioned buccally in the premolar/molar region.

The volunteers were randomly allocated into one of 3 groups: 5 mins erosion repeated x3, 10 mins erosion repeated x3 or 15 mins erosion repeated x3 and a coin was flipped to determine which side the samples were to be removed for ex vivo immersion with tails for left and heads for right. . At the beginning of the study visit the splints were inserted and worn for 30 minutes. Following which the enamel samples (1 polished and 1 unpolished) were removed from one side to begin the erosion regime. For in vivo erosion each participant was asked to rinse with orange juice for their either time 5, 10 or 15 minutes. This was standardised by setting up cups with 10 mL of the orange juice and a timer set at 1 minute. The participant was asked to insert the liquid into their mouths start the time and when the alarm sounded expectorate and repeat until they completed his/her time allocation of either 5, 10 or 15 minutes. Simultaneously the ex vivo samples were immersed in 20 mL of orange juice and agitated at 62 rpm for the allocated time using an orbital shaker (Stuart Scientific, Mini Orbital Shaker S05, Bibby). This completed one cycle after which the removed samples were reinserted into the splint which was worn for a further hour after which the rinsing/immersion regime was repeated. The process was repeated a further instance to complete 3 cycles of erosion. After the 3rd and final erosion cycle the participants were given a desensitising toothpaste Sensodyne Repair & Protect (GSK, Weybridge, UK).

The unpolished enamel samples were analysed before and after the experiment to measure changes in surface texture. Whereas, the polished samples were analysed for surface texture, hardness change and tissue loss.

ELIGIBILITY:
Inclusion Criteria:

* mild erosive tooth wear maximum score of 2 in each sextant and cumulative score no more than 8, aged 18 years and over, willing to participate, not enrolled in any other research, more than 20 anterior and posterior teeth, no active carious lesions and a maximum BPE score of 2 in one sextant (no periodontal disease).

Exclusion Criteria:

* pregnancy or breast feeding, medical history likely to impact on attendance or mobility, insulin dependent diabetes, saliva diagnoses (xerostomia), lower orthodontic appliances, dentine hypersensitivity, defective restoration of the occlusal or incisal surfaces of upper anterior teeth and first molars and any condition that precluded consumption of 300 ml of orange juice a day for 5 consecutive days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-05-29 (Actual)

PRIMARY OUTCOMES:
Microhardness (KHN) | 12 weeks
  To measure microhardness of enamel samples using a microhardness tester before and after the intervention. The units will be KHN

SECONDARY OUTCOMES:
Surface roughness | 12 weeks
  To measure surface roughness of enamel samples using anon contact profilometer before and after the intervention. The units will be microns.
Step height loss | 12 weeks
  To measure step height loss of enamel samples following the intervention using a non contact profilometer. The units will be microns.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mullan F, Austin RS, Parkinson CR, Bartlett DW. An in-situ pilot study to investigate the native clinical resistance of enamel to erosion. J Dent. 2018 Mar;70:124-128. doi: 10.1016/j.jdent.2018.01.005. Epub 2018 Jan 12. PMID 29339202